CLINICAL TRIAL: NCT02291536
Title: Processing of Salient Emotional Stimuli as a Function of Tetrahydrocannabinol (THC) and Cannabidiol (CBD)
Acronym: AB_THC_CBD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Institute of Mental Health, Mannheim (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: AB_THC_CBD
Record Dates: First submitted 2014-11-11; First posted 2014-11-14 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2014-11

CONDITIONS: Healthy Humans
Keywords: THC and CBD; Attentional blink
MeSH Terms: conditions — Color Vision Defects | interventions — Dronabinol; Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- tetrahydrocannabinol (Experimental): oral administration of 10mg of tetrahydrocannabinol, once
  Interventions: Drug: tetrahydrocannabinol
- cannabidiol (Experimental): oral administration of cannabidiol, 600mg, once
  Interventions: Drug: cannabidiol
- placebo (Placebo Comparator): oral administration of placebo, once
  Interventions: Other: placebo

INTERVENTIONS:
Drug: tetrahydrocannabinol
  Arms: tetrahydrocannabinol
Drug: cannabidiol
  Arms: cannabidiol
Other: placebo
  Arms: placebo

SUMMARY:
Attentional blink refers to a phenomenon where the detection of the second of two target stimuli that are presented in Short succession within a stream of stimuli is impaired. This is explained by an insufficient availability of attentional resources. Additionally, emotionally salient stimuli, like for example pictures with a positive or negative content, are detected more often compared to neutral pictures during this attentional blink period.

Cannabinoids are involved in the modulation of cognitive, attentional, and emotional processes. Interestingly, data from animals suggests that THC and CBD, both active ingredients in the Cannabis sativa plant, have opposing effects on brain cannabinoid (CB1) receptors. CB1 receptors modulate the expression of emotionally salient conditioned association in rats, if salience processes in humans are modulated in the same way remains unclear.

Employing a task to detect salient stimuli, Bhattacharyya et al. (2012) showed that THC seems to make non-salient standard stimuli more salient. They showed decreased activation of the right caudate and increased right prefrontal cortex stimuli during processing of salient stimuli. Importantly, this was associated with decreased response times to standard relative to oddball stimuli. Generally, THC and CBD differentially modulate brain areas associated with attentional salience processing. For example THC seems to increase prefrontal and striatal activation whereas CBD seems to decrease it.

The investigators assume that THC increases the number of correctly detected emotional stimuli during the attentional blink period, whereas CBD has no effect. Additionally, the investigators assume that pictures of the positive category are detected with higher accuracy than negative ones under the influence of THC.

ELIGIBILITY:
Inclusion Criteria:

* male
* age between 18 and 65 years
* right-handed

Exclusion Criteria:

* consumption of cannabis more than 5 times
* substance abuse (apart from nicotine)
* psychiatric disorders
* epilepsy
* chronic diseases (e.g. diabetes)

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Correctly identified emotional pictures during the attentional blink period | immediate
  Number of correctly identified emotional pictures that were presented during the attentional blink period.

SECONDARY OUTCOMES:
Reaction time to correctly identified emotional pictures during the attentional blink period | immediate
  Reaction time (in ms) of the button press to the correctly identified emotional pictures that were presented during the attentional blink period.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Grimm, MD, Principal Investigator — Central Institute of Mental Health, Mannheim
Locations (1):
- Central Institute of Mental Health, Mannheim, Germany